CLINICAL TRIAL: NCT00730730
Title: The Medtronic Complete® Self-Expanding Stent and Stent Delivery System Registry: a Non-randomized Prospective, Multicenter, Consecutive Registry
Brief Title: The Complete® Self-Expanding Stent and Stent Delivery System Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP084; IDE G070114
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-02

CONDITIONS: Peripheral Vascular Disease
Keywords: Iliac Artery, Peripheral Vascular Disease (PVD)
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Complete SE Iliac Stent (Experimental): Complete SE Iliac Stent
  Interventions: Device: Complete SE Iliac Stent

INTERVENTIONS:
Device: Complete SE Iliac Stent — Iliac stenting
Device: Complete SE Iliac Stent — Self-expanding stent

SUMMARY:
The purpose of this study is to show if a new delivery system with a modified stent is safe in treating occluded iliac arteries in patients with peripheral vascular disease. The modified Complete SE delivery system is hypothesized to assist physicians with more accurate stent placement reducing the likelihood of stent 'jumping' seen with the use of many self-expanding stent systems.

DETAILED DESCRIPTION:
The study is being conducted to collect the 30-day safety data on the stent delivery system for all subjects enrolled into the study (with a minimum of 50 subjects enrolled) as well as the long-term 9-month safety and efficacy data on all subjects enrolled (with a minimum of 10 subjects enrolled into the study having the 120mm length stent implanted).

ELIGIBILITY:
Inclusion Criteria:

* The lesion(s) is either de-novo or restenotic in nature, located in either the common iliac artery or the external iliac artery and is >50% stenosed
* Target vessel reference diameter ≥ 4.5 mm and ≤ 9.5 and can accommodate stent diameters of 6.0 - 10.0mm
* Subject is either asymptomatic with a lesion stenosis ≥70% or symptomatic with a lesion stenosis ≥50% with an Ankle Brachial Index (ABI) < 0.90 or Toe Brachial Index (TBI) <0.80 or an abnormal Pulse Volume Recording (PVR);
* Total lesion length is < 110 mm;

Exclusion Criteria:

* Excessive Peripheral Vascular Disease (PVD), unresolved fresh thrombus or tortuosity or a target lesion/vessel that is heavily calcified ;
* Tissue loss in the extremity: category 5 or 6 on the Rutherford scale;
* Target lesion has a previous stent, or is within a prosthetic vascular bypass graft or within 1 cm of a graft anastomosis;
* Target lesion is within an aneurysm or associated with an aneurysm in the vessel segment proximal or distal to the target lesion;
* Lesion requires treatment with a non-standard device associated with Percutaneous Transluminal Angioplasty (PTA) prior to stent placement;
* Inadequate distal run-off;
* Planned interventional procedure or vascular surgery to target vessel within 30 days pre- or post-index iliac procedure;
* History of bleeding diatheses or coagulopathy or will refuse blood transfusions;
* Platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or White Blood Count (WBC) <3,000 cells/mm3;
* Creatinine >2.0 mg/dl;
* Participation in another investigational device or drug study and has not completed the primary endpoint(s) follow-up phase of that study at least 30 days prior to enrollment in this trial or the subject has previously been enrolled in this Registry;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Molnar, MD, Principal Investigator — Michigan Vascular Research Center; William Gray, Principal Investigator — New York Presbyterian Hospital/Columbia Campus
Locations (2):
- United States (2):
  - Michigan Vascular Research Center, Flint, Michigan
  - New York Presbyterian Hospital, Columbia Campus, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Complete SE Iliac Stent: Iliac stenting (Complete® Self-Expanding Stent) for the treatment of de novo and restenotic lesions in iliac arteries in subjects with peripheral vascular disease (PVD)
Period: Overall Study
Arm/Group | Complete SE Iliac Stent
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Iliac Stenting: Iliac stenting (Complete® Self-Expanding Stent) for the treatment of de novo and restenotic lesions in iliac arteries in subjects with peripheral vascular disease (PVD)
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Major Adverse Events (MAE)
Description: Major adverse events (MAE) defined as any death, target limb loss or clinically-driven Target Lesion Revascularization (TLR)/Target Vessel Revascularization (TVR) with percutaneous transluminal angioplasty or aorto-iliac bypass graft) for all subjects enrolled into the registry
Time Frame: 30 days
Population: Intent-to-treat population (ITT)
Measure: Number; unit: participants
Arm/Group | Complete SE Iliac Stent
Number analyzed (Participants) | 50
participants | 0

2. Secondary Outcome: Number of Participants With Acute Success
Description: angiographic evidence of < 30 % final residual stenosis of the target lesion after stent placement with no occurrence of a device- related, procedure-related MAE or vascular event (stent thrombosis, major bleeding complications)
Time Frame: from after stent placement to prior to hospital discharge (up to 3 days)
Population: Intent to Treat population(ITT); missing angiographic data for one patient
Measure: Number; unit: participants
Arm/Group | Complete SE Iliac Stent
Number analyzed (Participants) | 49
participants | 44

3. Secondary Outcome: Number of Limbs With Improvement Using Rutherford Scale to Determine Clinical Success.
Description: Improvement of Rutherford scale by ≥ 1 category between pre-procedure (Baseline) and 30-day follow-up-
  * Category 0: Asymptomatic, no hemodynamically significant occlusive disease;
  * Category 1: Mild claudication;
  * Category 2: Moderate claudication;
  * Category 3: Severe claudication;
  * Category 4: Ischemic rest pain;
  * Category 5: Minor tissue loss; non-healing ulcer; focal gangrene with diffuse pedal ischemia;
  * Category 6: Major tissue loss extending above transmetatarsal level;functional foot no longer salvageable
Time Frame: From baseline up to 30-days
Population: Analysis calculated using number of evaluable limbs with Rutherford results; data missing for two limbs
Measure: Number; unit: limbs
Units Other Than Participants: limbs
Arm/Group | Complete SE Iliac Stent
Number analyzed (Participants) | 50
Number analyzed (limbs) | 54
limbs | 46

4. Secondary Outcome: Number of Limbs With Improvement Using Ankle-brachial Index and Toe Brachial Index to Determine Hemodynamic Success.
Description: Improvement in ankle-brachial index (ABI) or toe-brachial index (TBI) > 0.10 over pre-procedure level OR deterioration by ≤ 0.15 from first post-procedure exam OR pulse volume recording (PVR) distal to the target lesion treated maintained at ≥ 5 mm above pre-procedure tracing for those subjects with no pre-procedure ABI/TBI.
  An ABI ≥ 0.90 is considered normal.
Time Frame: From baseline up to 30-days
Population: Evaluable Ankle-brachial Index (ABI)/Toe brachial Index (TBI)result: missing data for 1 limb
Measure: Number; unit: limbs
Units Other Than Participants: limbs
Arm/Group | Complete SE Iliac Stent
Number analyzed (Participants) | 50
Number analyzed (limbs) | 55
limbs | 55 [93.5 to 100]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Iliac Stenting
Serious Adverse Events (participants affected / at risk) | 5/50
Other Adverse Events (participants affected / at risk) | 4/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iliac Stenting (N=50)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Dissection - Target Vessel (Vascular disorders) | 1 (1)
NSTEMI - Acute (Cardiac disorders) | 1 (1)
Pseudoaneurysm Left Femoral Artery (Injury, poisoning and procedural complications) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retroperitoneal Bleed (Gastrointestinal disorders) | 1 (1)
Right Lower Extremity Gangrene (Vascular disorders) | 1 (1)
Right Toe Gangrene (Vascular disorders) | 1 (1)
Shock Liver (Hepatobiliary disorders) | 1 (1)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iliac Stenting (N=50)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator/Institution agree to submit to Sponsor copies of any proposed publication/public presentation ("Proposed Publication") at least sixty (60) calendar days in advance of dissemination. Sponsor will review/comment within thirty (30) calendar days after receipt thereof. If Sponsor objects to dissemination of any part of the Proposed Publication, Investigator, and Institution shall refrain from disseminating or presenting such Proposed Publication until Sponsor is satisfied.